CLINICAL TRIAL: NCT00594295
Title: Follow-up of Bone Quality in Long-Term Bone Marrow Transplant Survivors
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-1098
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2010-04

CONDITIONS: Osteoporotic Fractures
MeSH Terms: conditions — Osteoporotic Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Brittle and broken bones can occur after organ transplantation. However, the long-term effects of bone marrow transplantation on bone health and the risk of breaking bones are not well understood. This study will help to assess how common it is for those who have received a bone marrow transplant to have fractures. It will also investigate blood tests related to bone health. This will be done by measuring bone mineral density and obtaining blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the initial "Assessment of skeletal status following allogeneic bone marrow transplantation" Study (HSC97-632-408).
* Able and willing to sign informed consent.

Exclusion Criteria:

* All of the contacted long-term BMT survivors that are willing to participate will be included in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Bone marrow transplant patients at least 6 years post transplant
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil C Binkley, MD, Principal Investigator — University of Wisconsin - Institute on Aging
Locations (1):
- University of Wisconsin Hospitals and Clinics, Madison, Wisconsin, United States